CLINICAL TRIAL: NCT01229670
Title: Effects of Aerobic Interval and Continuous Exercise Trainings on Cardiovascular Hemorheological Characteristics and Atherothrombosis/Angiogenesis-related Variables in Patients With Chronic Heart Failure
Brief Title: Effects of Aerobic Interval and Continuous Exercise Trainings in Patients With Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Chang Gung University (Other)
Responsible Party: Jong-Shyan Wang, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-3605B
Record Dates: First submitted 2010-10-18; First posted 2010-10-28 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Cardiac and Hemodynamic Response; Blood Flow Distribution and Oxygen Uptake Efficiency; Hemorheology Modulated by Erythrocyte; Atherothrombosis Modulated by Monocyte; Angiogenesis Modulated by EPC
Keywords: Heart failure; Hemorheology; Atherothrombosis; Angiogenesis
MeSH Terms: conditions — Heart Failure; Thrombosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aerobic intermittent group (Experimental): aerobic intermittent group
  Interventions: Other: exercise
- aerobic continuous group (Experimental): aerobic continuous group
  Interventions: Other: exercise
- control (No Intervention): home exercise group
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — * 1.exercise(Aerobic interval training (AIT)): training with 90% of VO2 peak and 40% of VO2 peak cycle for total 30 minutes exercise time
  * 2.exercise(moderate continuous training (MCT)):training with 60% of VO2peak for 30 min

SUMMARY:
Heart failure (HF) is a major and increasingly common cardiovascular syndrome, and is the end result of many cardiovascular disorders. It has been reported that HF patients with pharmacological therapy often remain burdened by dyspnea and fatigue, diminished exercise tolerance, reduced quality of life, recurrent hospitalizations, and early mortality. HF is associated with neurohumoral changes as the body attempts to reverse the effect of reduced cardiac output and organ perfusion. Persistent neurohumoral excitation, however, actually results in deterioration of myocardial function with inflammatory response, end-organ damage, and skeletal muscle derangement, which lead to worsened exercise capacity.

Physical training can have beneficial effects on neurohumoral, inflammatory, metabolic and central hemodynamic responses, as well as on endothelial, skeletal muscle and cardiovascular function, leading to improvement in functional capacity and quality of life. All these training-induced changes can effectively counteract the progression of deleterious compensatory mechanisms of HF.

Several lines of evidence suggest greater aerobic and cardiovascular adaptations after high-intensity exercise than with moderate levels in patients with coronary artery disease or left ventricular dysfunction function and in healthy subjects. Aerobic interval training (AIT) involving periods at 90% of VO2peak has been shown to rescue impaired cardiomyocyte contractility, attenuate myocardial hypertrophy, and reduce myocardial expression of atrial natriuretic peptide in animal model of post-infarction heart failure. However, underlying mechanisms of AIT-improved regulations remain unclear.

The different effects of AIT and moderate continuous training (MCT) on hemorheology, atherothrombosis or angiogenesis modulated by erythrocyte, monocyte or EPC in patients with CHF have been not investigated yet. Accordingly, the investigators will conduct this three-year study to clarify how the two exercise trainings affect cardiovascular hemorheological characteristics and atherothrombosis/ angiogenesis-related variables in patients with chronic heart failure. The investigators expect that these results obtained from this study can aid in determining appropriate exercise intervention to improve aerobic fitness as well as simultaneously improve hemodynamic control and minimize the risk of thrombogenesis in patients with CHF.

DETAILED DESCRIPTION:
Heart failure (HF) is a major and increasingly common cardiovascular syndrome, and is the end result of many cardiovascular disorders. It has been reported that HF patients with pharmacological therapy often remain burdened by dyspnea and fatigue, diminished exercise tolerance, reduced quality of life, recurrent hospitalizations, and early mortality. HF is associated with neurohumoral changes as the body attempts to reverse the effect of reduced cardiac output and organ perfusion. Persistent neurohumoral excitation, however, actually results in deterioration of myocardial function with inflammatory response, end-organ damage, and skeletal muscle derangement, which lead to worsened exercise capacity.

Physical training can have beneficial effects on neurohumoral, inflammatory, metabolic and central hemodynamic responses, as well as on endothelial, skeletal muscle and cardiovascular function, leading to improvement in functional capacity and quality of life. All these training-induced changes can effectively counteract the progression of deleterious compensatory mechanisms of HF. Which exercise intensity yields maximal beneficial adaptations is controversial.

Several lines of evidence suggest greater aerobic and cardiovascular adaptations after high-intensity exercise than with low and moderate levels in patients with coronary artery disease or left ventricular dysfunction function and in healthy subjects. Aerobic interval training (AIT) involving periods at 90% of VO2peak has been shown to rescue impaired cardiomyocyte contractility, attenuate myocardial hypertrophy, and reduce myocardial expression of atrial natriuretic peptide in animal model of post-infarction heart failure.

However, underlying mechanisms of AIT-improved regulations of cardiac hemodynamics and risk factors in patients with CHF remain unclear.

Pathological erythrocyte deformability and aggregation reduces capillary perfusion and oxygen transfer to tissue, resulting in tissue ischemia or infraction. Shedding of procoagulant-rich microparticles from activated monocytes can accelerate the pathogenesis of atherothrombosis. Bone marrow-derived, circulating endothelial progenitor cells (EPC) is contributes to the maintenance of endothelial function and organ perfusion by mechanisms ranging from endothelial repair to angiogenesis. However, the different effects of AIT and moderate continuous training (MCT) on hemorheology, atherothrombosis or angiogenesis modulated by erythrocyte, monocyte or EPC in patients with CHF have been not investigated yet.

Accordingly, we will conduct this three-year study that includes 1st year study: the effects of AIT and MCT on hemorheology modulated by erythrocyte in patients with CHF; 2nd year: the effects of AIT and MCT on atherothrombosis modulated by monocyte in patients with CHF; and 3rd year study: the effects of AIT and MCT on angiogenesis modulated by EPC in patients with CHF to clarify how the two exercise trainings affect cardiovascular hemorheological characteristics and atherothrombosis/ angiogenesis-related variables in patients with chronic heart failure. We expect that these results obtained from this study can aid in determining appropriate exercise intervention to improve aerobic fitness as well as simultaneously improve hemodynamic control and minimize the risk of thrombogenesis in patients with CHF.

ELIGIBILITY:
Inclusion Criteria:

* cardiac event with optimal medial treatment within 3 months and have 4 more weeks spared from heart disease attack or major cardiac procedure.

Exclusion Criteria:

* unstable angina pectoris,
* uncompensated heart failure,
* myocardial infarction during the past 4 weeks,
* complex ventricular arrhythmias,
* orthopedic or neurological limitations to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
ventilation efficacy | three year
  Ventilation efficacy could be show as ventilation equivalent(minute ventilation / oxygen consumption (VE/VO2) or minute ventilation / Carbon dioxide production (VE/VCO2). The slope of VE/VCO2 predict mortality in HF patient. These data ia available during cardiopulmonary exercise test(CPX or CPET). We also got other traditional data including Peak HR, Peak O2 consumption, Peak workload......

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Shyan Wang, Ph.D, Principal Investigator — Chamg Gung university
Locations (1):
- Chang Gung University, Kwei-Shan., Tao-Yuan, Taiwan

REFERENCES:
- [Background] Rognmo O, Hetland E, Helgerud J, Hoff J, Slordahl SA. High intensity aerobic interval exercise is superior to moderate intensity exercise for increasing aerobic capacity in patients with coronary artery disease. Eur J Cardiovasc Prev Rehabil. 2004 Jun;11(3):216-22. doi: 10.1097/01.hjr.0000131677.96762.0c. PMID 15179103
- [Background] Ribeiro JP, Stein R, Chiappa GR. Beyond peak oxygen uptake: new prognostic markers from gas exchange exercise tests in chronic heart failure. J Cardiopulm Rehabil. 2006 Mar-Apr;26(2):63-71. doi: 10.1097/00008483-200603000-00001. No abstract available. PMID 16569970
- [Background] Engoren M, Barbee D. Comparison of cardiac output determined by bioimpedance, thermodilution, and the Fick method. Am J Crit Care. 2005 Jan;14(1):40-5. PMID 15608107
- [Background] Belardinelli R, Barstow TJ, Porszasz J, Wasserman K. Changes in skeletal muscle oxygenation during incremental exercise measured with near infrared spectroscopy. Eur J Appl Physiol Occup Physiol. 1995;70(6):487-92. doi: 10.1007/BF00634377. PMID 7556120
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726